CLINICAL TRIAL: NCT01070940
Title: L-NMMA's Effect on Renal and Cardiovascular Variables in Healthy Subjects. A Randomized, Placebo-controlled Crossover Study.
Brief Title: L-NMMA Dose-response Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Thomas Larsen, M.D., Departments of Medical Research, Holstebro Hospital
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: EBP.FHC.1.2009; 2009-017001-11 (EudraCT Number)
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: L-NMMA; blood pressure; arterial stiffness; pulse wave velocity; augmentation index; dose-response; healthy subjects; GFR
MeSH Terms: interventions — omega-N-Methylarginine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Isotonic saline infusion (Placebo Comparator)
  Interventions: Drug: Placebo
- Intravenous L-NMMA dose 2 (Active Comparator)
  Interventions: Drug: NG-monomethyl-L-arginine (L-NMMA)
- Intravenous L-NMMA dose 3 (Active Comparator)
  Interventions: Drug: NG-monomethyl-L-arginine (L-NMMA)
- Intravenous L-NMMA dose 1 (Active Comparator)
  Interventions: Drug: NG-monomethyl-L-arginine (L-NMMA)

INTERVENTIONS:
Drug: NG-monomethyl-L-arginine (L-NMMA) — 3 mg/kg IV priming dose + 2 mg/kg/hr IV infusion for 1 hour
  Arms: Intravenous L-NMMA dose 1
Drug: NG-monomethyl-L-arginine (L-NMMA) — 6 mg/kg IV priming dose + 4 mg/kg/hr IV infusion for 1 hour
  Arms: Intravenous L-NMMA dose 3
Drug: NG-monomethyl-L-arginine (L-NMMA) — 4.5 mg/kg IV priming dose + 3 mg/kg/hr IV infusion for 1 hour
  Arms: Intravenous L-NMMA dose 2
Drug: Placebo — Isotonic saline solution IV priming dose + IV infusion for 1 hour
  Arms: Isotonic saline infusion

SUMMARY:
The purpose of this study is to investigate the effect of different levels of nitric oxide inhibition on blood pressure and arterial stiffness in healthy subjects. L-NMMA, an inhibitor of the nitric oxide synthase, is administered as bolus injection followed by continuous infusion, and is expected to raise blood pressure and arterial stiffness according to L-NMMA dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 18-35 years
* BMI 18.5-30.0

Exclusion Criteria:

* Tobacco or illicit drug use
* Current use of any prescription or non-prescription drugs
* Alcohol abuse
* History of heart failure, lever failure, chronic kidney disease or cerebral insult
* Diabetes
* Clinical or paraclinical signs of infection
* Pathologic ECG
* Ambulatory blood pressure >140/90 mmHg
* Abnormal blood or urin screening tests

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 6 hours

SECONDARY OUTCOMES:
GFR | 6 hours
Arterial Stiffness | 6 hours
Fractional excretion of sodium | 6 hours
Fractional excretion of potassium | 6 hours
Plasma renin concentration | 6 hour
Plasma angiotensin II | 6 hours
Plasma aldosterone | 6 hour

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Larsen, M.D., Principal Investigator — Departments of Medical Research, Holstebro Hospital; Frank H Christensen, M.D., Principal Investigator — Departments of Medical Research, Holstebro Hospital; Erling B Pedersen, Dr.med., Principal Investigator — Departments of Medical Research, Holstebro Hospital; Jesper N Bech, Ph.d., Principal Investigator — Departments of Medical Research, Holstebro Hospital
Locations (1):
- Departments of Medical Research, Holstebro, Holstebro, Denmark